CLINICAL TRIAL: NCT02202694
Title: Feasibility Study of Culturally Adapted Cognitive Behavior Therapy for Psychosis in Pakistan
Brief Title: Culturally Adapted Cognitive Behavior Therapy for Psychosis in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other); Dow University of Health Sciences (Other); Abbasi Shaheed Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT-PSY-01
Record Dates: First submitted 2014-04-15; First posted 2014-07-29 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2014-07

CONDITIONS: Psychosis
Keywords: CBT, Psychosis, cultural adaptation, Pakistan
MeSH Terms: conditions — Psychotic Disorders; Color Vision Defects | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Culturally Adapted Cognitive Behavior Therapy
  Interventions: Behavioral: Culturally Adapted Cognitive behavior therapy
- Control (No Intervention): Patients who will be randomized to the "treatment as usual" arm will receive routine care

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive behavior therapy — This 12 session Multimodal Psychosocial Intervention will include a supportive component, an educational component, psychosocial component
  Other Names: Psychosocial intervention
  Arms: Intervention

SUMMARY:
Aim:

To assess the feasibility of application of culturally-adapted CBT (CaCBTp) for use in Pakistan.

Design:

Randomized Control Trial

Setting:

Psychiatry Departments of General Hospitals in Karachi.

Participants:

A total of 36 patients with a diagnosis of psychotic disorder will be randomized to a psychological intervention or treatment as usual arm.

Intervention:

Culturally Adapted Cognitive Behavioral Therapy (CBT)

Outcome measure:

Positive and Negative syndrome scale (PANSS) Psychotic symptoms Rating Scales (PSYRATS)

DETAILED DESCRIPTION:
The purpose of the study is to test the feasibility of culturally adaptive CBT for Psychosis in Pakistan

Primary :

-To assess the feasibility of application of culturally-adapted CBT (CaCBTp) for use in Pakistan.

Secondary:

* To assess fidelity of culturally-adapted CBT for psychosis.
* To further modify CaCBTp in accordance with findings of feasibility study

The Participants will be recruited from psychiatric department of different hospitals.They will be randomly divided into two groups; intervention group and treatment-as-usual group. A total of thirtysix participants will be recruited in the feasibility study and divided equally into two arms. This will ensure that, even after loss to follow-up, the investigators will have at least 12 subjects per group for analysis (FDA guidance http://www.fda.gov/cder/guidance/5356fnl.pdf. Randomization will be carried out by the on offsite statistician . This will provide a reliable geographically remote service. For intervention group twelve sessions of CaCBTp will be delivered by trained research clinician for a period of three months. Participants in the treatment as usual (TAU) group will be given details of intervention at the end of the study and interested Participants will be offered CaCBTp.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Psychosis established by clinician using ICD10 criteria.
2. Individuals aged between 18-65.
3. Should not have learning disability.
4. Resident of Karachi.
5. Participant is able to give informed written consent

Exclusion Criteria:

1. Severe illness which may affect capacity or markedly affect their ability to participate in interview, e.g. very thought disordered or distressed by symptoms.
2. Severe drug or alcohol problem (i.e., those who fulfill the criteria for dependence according to ICD10 RDC).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Positive and Negative syndrome scale (PANSS) | up to 6 months
  The PANSS is a structured clinical interview consisting of 30 items designed to assess severity of symptoms over the past week on a 7-point scale.

SECONDARY OUTCOMES:
Psychotic Symptom Rating Scales (PSYRATS) | Baseline ,3 months & 6 months
  The PSYRATS consists of 17 items that focus on auditory hallucinations and delusions experienced over the past week.
Insight rating scale | Baseline ,3 months & 6 months
  Assesses Improvement in insight
Calgary Depression Scale for Schizophrenia | Baseline ,3 months & 6 months
  This is a nine-item scale developed by Addington et al. to assess depression in schizophrenia.
Short Explanatory Model Interview | Baseline ,3 months & 6 months
  used to elicit beliefs of mental illness

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, MD, Principal Investigator — Pakistan Institute of Learning and Living, University of Manchester; Imran Chaudhry, MD, Principal Investigator — University of Manchester; Farooq Naeem, MRCPsych, Principal Investigator — Pakistan Institute of Learning and Living, University of Southampton; Raza ur Rehman, FCPS, Principal Investigator — Dow University of Health Sciences; Ajmal Kazmi, Principal Investigator — Pakistan Institute of Living and Learning; Munir Hamirani, FCPS, Principal Investigator — Abbasi Shaheed Hospital
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Husain MO, Chaudhry IB, Mehmood N, Rehman RU, Kazmi A, Hamirani M, Kiran T, Bukhsh A, Bassett P, Husain MI, Naeem F, Husain N. Pilot randomised controlled trial of culturally adapted cognitive behavior therapy for psychosis (CaCBTp) in Pakistan. BMC Health Serv Res. 2017 Dec 6;17(1):808. doi: 10.1186/s12913-017-2740-z. PMID 29207980